CLINICAL TRIAL: NCT01476696
Title: An Open-Label, Dose-Ranging Study of Prasugrel in Pediatric Patients With Sickle Cell Disease
Brief Title: A Study of Prasugrel in Pediatric Participants With Sickle Cell Disease
Acronym: Crescent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12324; H7T-MC-TACX (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; pediatrics; SCD; children; child; kids; pain crisis; sickle cell anemia; sickle cell pain
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Prasugrel Single Dose (Experimental): Prasugrel 0.03 milligrams per kilogram (mg/kg) to 0.60 mg/kg dosage to be titrated up or down based on desired platelet inhibition, administered orally [oral-disintegrating tablet (ODT)], single dose given up to 3 occasions, at different strengths, with up to 18 days between doses.
  Interventions: Drug: Prasugrel
- Part B: Prasugrel Once-Daily Dose (Experimental): Daily prasugrel dose (mg/kg) that is expected to achieve mean platelet activation inhibition of 30% administered orally, once daily for 10-18 days and then followed by prasugrel dose (mg/kg) that is expected to achieve mean platelet activation inhibition of 50% administered orally, once daily for 10-18 days, for a total of 20-36 days.
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Administered orally
  Other Names: Effient; Efient; LY640315; CS-747

SUMMARY:
The purpose of this study is to determine the correct prasugrel dosage to be given to children with sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Are male or female with SCD [(homozygous sickle cell (HbSS) and hemoglobin S beta ^0 thalassemia (HbS β^0 thalassemia)]
* Have a body weight ≥12 kilograms (kg) and are ≥2 to <18 years of age at the time of screening
* If participants are ≥2 and ≤16 years of age, have had a transcranial Doppler within the last year
* Participants on hydroxyurea must be on a stable dose for the 60 days prior to enrollment without signs of hematologic toxicity at screening
* Have a legal representative that is in competent mental condition to provide written informed consent on behalf of the study participant before entering the study. The child may be required to give documented assent, if required by local regulations.
* If sexually active, has a negative pregnancy test at screening (if female) and agrees to use a reliable method of birth control during the study (for both males and females)

Exclusion Criteria:

* Known to have hemoglobin C sickle cell (HbSC) or hemoglobin S beta ^plus thalassemia (HbS β^+ thalassemia) genotypes
* Vaso-occlusive crisis (VOC) requiring medical attention within 15 days prior to screening
* Have a concomitant medical illness (for example, terminal malignancy) that in the opinion of the investigator is associated with reduced survival
* Hepatic dysfunction characterized by alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal (ULN)
* Renal dysfunction requiring chronic dialysis or creatinine ≥ 1.5 milligrams per deciliter (mg/dL)
* Contraindication for antiplatelet therapy
* History of intolerance or allergy to approved thienopyridines (clopidogrel, ticlopidine, or prasugrel)
* Participants with a hematocrit <18%
* History of abnormal or conditional transcranial Doppler [velocity in middle cerebral or carotid artery ≥170 centimeters per second (cm/sec)] within the last year
* Any history of bleeding diathesis
* Any history of renal papillary necrosis
* Active internal bleeding
* History of spontaneous gastrointestinal bleeding
* Gross hematuria or > 300 red blood cells (RBC)/high-powered field (HPF) on urinalysis at the time of screening
* Any history of vitreous hemorrhage
* Prior history of hemorrhagic or ischemic stroke, a transient ischemic attack (TIA), or other intracranial hemorrhage
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding
* Platelet count <100,000 per microliter (μl) of blood
* Have had recent surgery (within 30 days prior to screening) or are scheduled to undergo surgery within the next 60 days
* History of dysfunctional uteral bleeding, in the judgment of the investigator
* Treatment with packed RBC or whole blood transfusion therapy within 30 days prior to dosing
* Any nonsteroidal anti-inflammatory drug (NSAID) use within 5 days prior to screening
* Any aspirin, warfarin, thienopyridine, or other antiplatelet medication use within 10 days prior to dosing
* Anticipated use of aspirin, warfarin, thienopyridine, or other antiplatelet medication during the study period

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC-GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts: Part A (single-dose range finding phase) then Part B (once-daily repeated dosing phase). Participants completing Part A could, but were not required to, participate in Part B. There were 2 dosing periods during Part B of the study.
Groups:
- Part A: Prasugrel Single Dose: Participants who only enrolled in Part A of the study.
  Part A: 0.03 milligrams per kilogram (mg/kg) up to 0.60 mg/kg Prasugrel, each dose titrated up or down for each participant in order to achieve desired platelet inhibition (20% to 50%). Single dose administered orally [oral-disintegrating tablet (ODT)] up to 3 times, at different mg/kg doses, with up to 18 days between doses.
- Part B: Prasugrel Once-Daily Dose: Participants who only enrolled in Part B of the study.
  Part B: Daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period during Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then pharmacodynamic (PD) response measured 4 hours later. Based on 4-hour PD response, each participant assigned to either 0.08 or 0.06 mg/kg Prasugrel, administered orally, once daily for the remainder of the first dosing period in Part B. For the second continuous 14 ± 4-day period, participants were administered 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on their steady-state PD response at the end of the first dosing period, such that the second dose would be unlikely to exceed 50% platelet inhibition. Participants received study drug for a total of 28 ± 8 days during Part B of the study.
- Part A Then Part B: Prasugrel Single Dose Then Once-Daily Dose: Participants who enrolled in Part A and B of study. Part A: 0.03 up to 0.60 mg/kg Prasugrel, each dose titrated up or down for each participant to achieve desired platelet inhibition (20% to 50%). Single dose administered orally, ODT, up to 3 times, at different mg/kg doses, with up to 18 days between doses.
  Part B: Daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period in Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then PD response measured 4 hours later. Based on 4-hour PD response, each participant assigned to 0.08 or 0.06 mg/kg Prasugrel once daily for remainder of first dosing period. For second 14 ± 4-day period, participants assigned to 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on steady-state PD response at end of first dosing period, such that the second dose would be unlikely to exceed 50% platelet inhibition.
Period: Overall Study
Arm/Group | Part A: Prasugrel Single Dose | Part B: Prasugrel Once-Daily Dose | Part A Then Part B: Prasugrel Single Dose Then Once-Daily Dose
Started | 15 | 9 | 9
Received at Least 1 Dose of Study Drug | 15 | 9 | 9
Completed | 12 | 8 | 9
Not Completed | 3 | 1 | 0
Not completed — Sponsor decision | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Entire Study Population: Participants enrolled in Part A, Part A and B, or only Part B of study. Part A: 0.03 up to 0.60 mg/kg Prasugrel, each dose titrated up or down for each participant to achieve desired platelet inhibition (20% to 50%). Single dose administered orally, ODT, up to 3 times, at different mg/kg doses, with up to 18 days between doses.
  Part B: Daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period in Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then PD response measured 4 hours later. Based on 4-hour PD response, each participant assigned to 0.08 or 0.06 mg/kg Prasugrel once daily for remainder of first dosing period. For second 14 ± 4-day period, participants assigned to 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on steady-state PD response at end of first dosing period, so that the second dose would be unlikely to exceed 50% platelet inhibition.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 33
Age, Customized [Number; unit: participants]
  ≥2 and ≤5 years | 7
  ≥6 and ≤11 years | 14
  ≥12 and ≤17 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 32
Region of Enrollment [Number; unit: participants]
  United States | 33
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 139.21 (22.663)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 38.55 (18.785)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 18.64 (4.091)
Genotype [Number; unit: participants] — The number of participants who have the homozygous sickle cell (HbSS) or hemoglobin S beta^0 thalassemia (HbS β^0 thalassemia)] sickle cell genotype.
  participants
    HbSS | 30
    HbS Beta^0 Thalassemia | 3

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Prasugrel Active Metabolite (Pras-AM)
Description: AUC of Pras-AM from time 0 up to the last sampling time of 4 hours postdose [AUC(0-tlast)] is reported by dose administered [0.03, 0.05, 0.07, 0.09, 0.11, 0.13, 0.15, 0.2, 0.25, 0.3, 0.35, 0.4, 0.45, 0.5, 0.55, and 0.6 milligrams per kilogram (mg/kg)] during Part A (single-dose range finding phase) and is reported for doses administered on site (0.06, 0.08, and 0.12 mg/kg) during Part B (once-daily repeated dosing phase) of the study. Four participants received the same dose at multiple visits where pharmacokinetic samples were collected.
Time Frame: Parts A and B: 0.5, 1, 1.5, 2, 4 hours postdose
Population: Participants who received at least 1 dose of prasugrel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 33
nanograms*hour per milliliter (ng*hr/mL)
  Part A: 0.03 mg/kg (n=2) | 8.68 (36)
  Part A: 0.05 mg/kg (n=2) | 14.5 (44)
  Part A: 0.07 mg/kg (n=2) | 20.8 (31)
  Part A: 0.09 mg/kg (n=2) | 31.3 (25)
  Part A: 0.11 mg/kg (n=1) | 22.2 (NA) — The geometric coefficient of variation could not be determined because data for only 1 profile were analyzed.
  Part A: 0.13 mg/kg (n=2) | 50.3 (20)
  Part A: 0.15 mg/kg (n=2) | 35.2 (86)
  Part A: 0.2 mg/kg (n=2) | 43.7 (48)
  Part A: 0.25 mg/kg (n=3) | 60.7 (88)
  Part A: 0.3 mg/kg (n=6) | 87.9 (52)
  Part A: 0.35 mg/kg (n=11) | 111 (59)
  Part A: 0.4 mg/kg (n=14) | 108 (55)
  Part A: 0.45 mg/kg (n=8) | 136 (53)
  Part A: 0.5 mg/kg (n=7) | 186 (36)
  Part A: 0.55 mg/kg (n=1) | 87.0 (NA) — The geometric coefficient of variation could not be determined because data for only 1 profile were analyzed.
  Part A: 0.6 mg/kg (n=3) | 299 (4)
  Part B: 0.06 mg/kg (n=7) | 16.3 (50)
  Part B: 0.08 mg/kg (n=17) | 27.1 (20)
  Part B: 0.12 mg/kg (n=8) | 38.5 (15)

2. Primary Outcome: Percentage of Platelet Inhibition as Measured by VerifyNow™P2Y12 (VN)
Description: Accumetrics VN assay: A point-of-care device that measures platelet aggregation. Percentage of platelet inhibition is reported by dose administered [0.03, 0.05, 0.07, 0.09, 0.11, 0.13, 0.15, 0.2, 0.25, 0.3, 0.35, 0.4, 0.45, 0.5, 0.55, and 0.6 milligrams per kilogram (mg/kg)] during Part A (single-dose range finding phase) and also during the once-daily repeated dosing phase in Part B, at steady state, 14 ± 4 days after each new dose (0.06, 0.08, and 0.12 mg/kg) is administered. One participant received the same dose at multiple visits (Part A) and one participant received the same daily dose during both dosing periods in Part B.
Time Frame: Part A: 4 hours postdose and Part B: at steady state (14 ± 4 days after the start of each new dosage)
Population: Participants who received at least 1 dose of prasugrel.
Measure: Mean (Standard Deviation); unit: percentage of platelet inhibition
Arm/Group | Entire Study Population
Number analyzed (Participants) | 33
percentage of platelet inhibition
  Part A: 0.03 mg/kg (n=2) | 2.0 (2.83)
  Part A: 0.05 mg/kg (n=2) | 0.0 (0.00)
  Part A: 0.07 mg/kg (n=2) | 0.0 (0.00)
  Part A: 0.08 mg/kg (n=18) | 7.7 (9.35)
  Part A: 0.09 mg/kg (n=2) | 2.5 (3.54)
  Part A: 0.11 mg/kg (n=1) | 0.0 (NA) — Could not be determined because data for only 1 participant were analyzed.
  Part A: 0.13 mg/kg (n=2) | 9.5 (13.44)
  Part A: 0.15 mg/kg (n=2) | 4.0 (0.00)
  Part A: 0.2 mg/kg (n=2) | 0.0 (0.00)
  Part A: 0.25 mg/kg (n=3) | 18.0 (18.52)
  Part A: 0.3 mg/kg (n=6) | 42.3 (27.21)
  Part A: 0.35 mg/kg (n=11) | 38.0 (28.46)
  Part A: 0.4 mg/kg (n=14) | 39.1 (26.77)
  Part A: 0.45 mg/kg (n=8) | 35.3 (27.16)
  Part A: 0.5 mg/kg (n=7) | 55.9 (27.85)
  Part A: 0.55 mg/kg (n=1) | 31.0 (NA) — Could not be determined because data for only 1 participant were analyzed.
  Part A: 0.6 mg/kg (n=3) | 70.3 (19.22)
  Part B: 0.06 mg/kg (n=8) | 38.6 (21.07)
  Part B: 0.08 mg/kg (n=18) | 37.8 (25.86)
  Part B: 0.12 mg/kg (n=8) | 48.1 (11.29)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Prasugrel Inactive Metabolite
Description: AUC of prasugrel inactive metabolite(s) from time 0 up to the last sampling time of 4 hours postdose [AUC(0-tlast)]. Improvements in bioanalytical methodology enabled direct measurement of Pras-AM from plasma, obviating the need to estimate its concentration from inactive downstream metabolite(s). Thus, the AUC of prasugrel inactive metabolite(s) was not analyzed.
Time Frame: Part A: 0.5, 1, 1.5, 2, 4 hours postdose
Population: No participants were analyzed.
Groups:
- Part A: Prasugrel Single Dose: Part A of the study: 0.03 up to 0.60 milligrams per kilogram (mg/kg) Prasugrel, each dose titrated up or down for each participant in order to achieve desired platelet inhibition (20% to 50%). Single dose administered orally [oral-disintegrating tablet (ODT)] up to 3 times, at different mg/kg doses, with up to 18 days between doses.
Arm/Group | Part A: Prasugrel Single Dose
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Pain
Description: The number of participants who answered "yes" to the first question in the Sickle Cell Disease Pain (SCD) Questionnaire is reported. Question 1: In the past 2 weeks, did you experience any sickle cell pain?
Time Frame: Part B: Baseline and Day14 ± 4 days postdose in each dosing period
Population: Participants who responded to Question 1 of the SCD Questionnaire. A participant could be counted more than once because there were 2 dosing periods during Part B of the study.
Measure: Number; unit: participants
Groups:
- Part B: Baseline: Participants in Part B of the study, prior to receiving treatment (Prasugrel once-daily doses).
- Part B: Prasugrel Once-Daily Dose (0.06 mg/kg): Participants who received 0.06 mg/kg Prasugrel administered orally, ODT, once daily, anytime (first or second dosing period) during Part B of the study, for a total of up to 36 days.
- Part B: Prasugrel Once-Daily Dose (0.08 mg/kg): Participants who received 0.08 mg/kg Prasugrel administered orally, ODT, once daily, anytime (first or second dosing period) during Part B of the study, for a total of up to 36 days.
- Part B: Prasugrel Once-Daily Dose (0.12 mg/kg): Participants who received 0.12 mg/kg Prasugrel administered orally, ODT, once daily, anytime (first or second dosing period) during Part B of the study, for a total of up to 36 days.
Arm/Group | Part B: Baseline | Part B: Prasugrel Once-Daily Dose (0.06 mg/kg) | Part B: Prasugrel Once-Daily Dose (0.08 mg/kg) | Part B: Prasugrel Once-Daily Dose (0.12 mg/kg)
Number analyzed (Participants) | 18 | 9 | 17 | 8
participants | 6 | 4 | 1 | 2

5. Secondary Outcome: Number of Participants With Hemorrhagic Events Requiring Medical Intervention
Description: Hemorrhagic events were determined by the study investigator. Medical intervention was defined as any medical attention resulting in therapy or further investigation, as determined by a trained medical professional.
Time Frame: Part B: Baseline up to Day 36
Population: Participants who received at least 1 dose of prasugrel.
Measure: Number; unit: participants
Groups:
- Part B: Prasugrel Once-Daily Dose: Part B: daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period during Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then pharmacodynamic (PD) response measured 4 hours later. Based on 4-hour PD response, each participant assigned to either 0.08 or 0.06 mg/kg Prasugrel administered orally, once daily for the remainder of the first dosing period in Part B. For the second continuous 14 ± 4-day period, participants were administered 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on their steady-state PD response at the end of the first dosing period, such that the second dose would be unlikely to exceed 50% platelet inhibition. Participants received study drug for a total of 28 ± 8 days during Part B of the study.
Arm/Group | Part B: Prasugrel Once-Daily Dose
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Groups:
- Part B: Prasugrel Once-Daily Dose: Participants who only enrolled in Part B of the study.
  Part B: Daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period during Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then pharmacodynamic (PD) response measured 4 hours later. Based on 4-hour PD response, each participant assigned to either 0.08 or 0.06 mg/kg Prasugrel administered orally, once daily for the remainder of the first dosing period in Part B. For the second continuous 14 ± 4-day period, participants were administered 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on their steady-state PD response at the end of the first dosing period, such that the second dose would be unlikely to exceed 50% platelet inhibition. Participants received study drug for a total of 28 ± 8 days during Part B of the study.
- Part A and Part B Participants: During Part A: Events reported during Part A for those participants who enrolled in Part A and Part B of study.
  Part A: 0.03 mg/kg up to 0.60 mg/kg Prasugrel, each dose titrated up or down for each participant in order to achieve desired platelet inhibition (20% to 50%). Single dose administered orally, ODT, up to 3 times, at different mg/kg doses, with up to 18 days between doses.
- Part A and Part B Participants: During Part B: Events reported during Part B for those participants who enrolled in Part A and Part B of study.
  Part B: Daily Prasugrel dose (mg/kg) expected to achieve mean platelet activation inhibition of 30%, administered orally, ODT, once daily for 14 ± 4 days (first dosing period during Part B). Initial dose, 0.08 mg/kg Prasugrel, administered then pharmacodynamic (PD) response measured 4 hours later. Based on 4-hour PD response, each participant assigned to either 0.08 or 0.06 mg/kg Prasugrel administered orally, once daily for the remainder of the first dosing period in Part B. For the second continuous 14 ± 4-day period, participants were administered 1 of 3 possible doses: 0.06, 0.08, or 0.12 mg/kg depending on their steady-state PD response at the end of the first dosing period, such that the second dose would be unlikely to exceed 50% platelet inhibition. Participants received study drug for a total of 28 ± 8 days during Part B of the study.
Arm/Group | Part A: Prasugrel Single Dose | Part B: Prasugrel Once-Daily Dose | Part A and Part B Participants: During Part A | Part A and Part B Participants: During Part B
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/15 | 4/9 | 6/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Prasugrel Single Dose (N=15) | Part B: Prasugrel Once-Daily Dose (N=9) | Part A and Part B Participants: During Part A (N=9) | Part A and Part B Participants: During Part B (N=9)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Prasugrel Single Dose (N=15) | Part B: Prasugrel Once-Daily Dose (N=9) | Part A and Part B Participants: During Part A (N=9) | Part A and Part B Participants: During Part B (N=9)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid bleeding (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/6 (0) | 1/4 (1) | 0/4 (0) | 0/4 (0)
Penis disorder (Reproductive system and breast disorders) | 0/6 (0) | 0/4 (0) | 1/4 (1) | 0/4 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Data for the Primary Outcome Measures 1 and 2 were collected for presentation of results in a scatter plot and were not intended to be summarized due to the limited number of participants per treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days